CLINICAL TRIAL: NCT07373873
Title: Assessment of Growth in Children With Congenital Heart Disease in Assuit University Children Hospital
Brief Title: Growth in Infants With Congenital Heart Disease at AUCH
Acronym: CHD-Growth
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lamia Mohammed Hussain Mohammed, Resident Doctor at Al-Mabrah Hospital, Assiut University
Other Study IDs: FMASU-PED-CHD-Growth-001
Record Dates: First submitted 2026-01-16; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Congenital Heart Disease (CHD)
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CHD Group: Infants and children aged 1 month to 2 years who were diagnosed with congenital heart disease (CHD) by echocardiography at Assiut University Children Hospital. This is a retrospective cohort; data on anthropometric measurements (weight, height/length, head circumference), type of CHD (cyanotic vs. acyanotic), and clinical history are collected from existing medical records. The growth parameters of this cohort will be compared against standard WHO or Egyptian growth reference charts to assess the impact of CHD on somatic growth.

SUMMARY:
Children with congenital heart disease (CHD) often experience growth problems. This study aims to assess and compare the growth (weight, height, head circumference) of infants and children with CHD against the expected growth standards for healthy children. This is a retrospective study that will review the medical records of children aged 1 month to 2 years who were diagnosed with CHD at Assiut University Children Hospital. The study will help understand how different types of CHD affect a child's growth, which is important for improving their nutritional care and overall management.

DETAILED DESCRIPTION:
Background:

Congenital heart disease (CHD) is the most common type of congenital anomaly and a leading cause of morbidity in children. Despite advances in medical and surgical care, growth retardation remains a frequent comorbidity in this population. The pathophysiology of growth failure differs between cyanotic and acyanotic CHD, involving factors such as chronic hypoxemia, increased metabolic demands, feeding difficulties, and congestive heart failure. A detailed assessment of growth patterns in children with CHD is crucial for optimizing nutritional interventions, determining the timing of surgical repair, and improving long-term outcomes.

Objective:

The primary objective of this study is to define the impact of congenital heart disease on the somatic growth of infants and children. This will be achieved by comparing anthropometric parameters (weight, height/length, and head circumference) of patients with CHD to established growth standards for healthy children.

Study Design:

This is a retrospective, comparative cohort study. Data will be collected from the existing medical records of patients followed at the Pediatric Cardiology Unit of Assiut University Children Hospital.

Participants:

The study group will include children aged 1 month to 2 years who have been diagnosed with CHD by echocardiography. Patients with known genetic syndromes (e.g., Down syndrome), major extracardiac anomalies, pre-existing endocrine or metabolic disorders affecting growth, preterm birth history, or those who have already undergone surgical or interventional procedures for their CHD will be excluded.

Methods:

For each eligible child, the following data will be extracted from the medical records:

Demographic Information: Age, sex, and residence.

Anthropometric Measurements: Weight, height/length, and head circumference recorded during hospital visits.

Clinical Data: Specific type of CHD (classified as cyanotic or acyanotic), history of hospitalizations, and other relevant clinical notes.

Growth Assessment: Anthropometric data will be assessed at key age points (6, 12, and 18 months) where available.

Statistical Analysis:

Data analysis will be performed using SPSS version 26. Continuous variables will be presented as mean ± standard deviation, and categorical variables as frequencies and percentages. Growth parameters of the CHD cohort will be compared to standard population norms using appropriate statistical tests (e.g., one-sample t-test). Comparisons between cyanotic and acyanotic groups will be conducted using independent samples t-test or Mann-Whitney U test, as applicable. A p-value of less than 0.05 will be considered statistically significant.

Ethical Considerations:

The study protocol has been approved by the Ethics of Scientific Research Committee, Faculty of Medicine, Assiut University. The research involves the analysis of existing, anonymized data from medical records.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 month to 2 years.
* Diagnosis of congenital heart disease (CHD) confirmed by echocardiography.
* Availability of anthropometric data in the medical record.

Exclusion Criteria:

* Presence of a known genetic syndrome or major extracardiac anomalies.
* Pre-existing endocrine or metabolic disorder affecting growth.
* Preterm birth (gestational age <37 weeks).
* Previous surgical/interventional procedure for CHD.

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — The study involves analysis of existing medical records. Eligibility for data inclusion is based on the biological sex (male or female) recorded in the patient's file at the time of clinical care, as growth reference standards are sex-specific. The study does not involve prospective recruitment where self-identified gender would be assessed.
Study Population: The study population consists of infants and young children (aged 1 month to 2 years) who were diagnosed with congenital heart disease (CHD) by echocardiography and were followed at the Pediatric Cardiology Unit of Assiut University Children Hospital. This is a retrospective cohort; participants are identified through a review of existing hospital medical records. The population includes patients with various types of CHD (both cyanotic and acyanotic) who have not yet undergone corrective cardiac surgery or intervention.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Weight-for-age z-score in children with congenital heart disease | At study enrollment (data extracted from medical records for age points 6, 12, and 18 months where available).
  Comparison of the mean weight-for-age z-score in children with congenital heart disease (CHD) against the standard population mean (z-score = 0) using WHO or Egyptian growth reference charts.

CONTACTS AND LOCATIONS:
Overall Officials: Emad-Eldeen Mahmoud Hammad mo Hammad, prof, Study Director — Assiut University
Locations (2):
- Egypt (2):
  - Assuit University Children Hospital - Cardiology Department, Asyut
  - Assuit University Children Hospital, Asyut

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) that underlie the published aggregated results will not be publicly deposited due to patient confidentiality and institutional data policies. However, de-identified data may be made available to qualified researchers upon reasonable request, subject to review and approval by the principal investigator and the Ethics Committee of Assiut University Faculty of Medicine. Requestors will need to provide a methodologically sound proposal and sign a data use agreement